CLINICAL TRIAL: NCT02183935
Title: Treatment of Morbidly Obese Adolescent With a Duodena-jejunal Liner - a Study on Efficacy and Pathophysiologic Mechanisms
Brief Title: Treatment of Morbidly Obese Adolescent With a Duodena-jejunal Liner
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Tadej Battelino, Prof. Dr., University Medical Centre Ljubljana
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EB-AD-39/03/14
Record Dates: First submitted 2014-06-30; First posted 2014-07-08 (Estimated); Last update posted 2020-07-10 (Actual); Status verified 2020-07

CONDITIONS: Obesity; Diabetes; Metabolic Syndrome
Keywords: Obesity; Diabetes; Metabolic syndrome; Gut hormones; Adipokines; Appetite; Adolescent
MeSH Terms: conditions — Obesity; Diabetes Mellitus; Metabolic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lifestyle counseling, metformin (No Intervention): Age, gender and BMI matched controls will be managed by lifestyle counseling and metformin if indicated.
- Duodeno - jejunal liner (Active Comparator): Duodeno-jejunal liner (Endobarrier) will be implanted for the duration of 12 months. During this time subjects will be regularly monitored for investigated parameters. In addition, subjects will be carefully monitored upon device removal for additional 12 months.
  Interventions: Device: Duodena-jejunal liner

INTERVENTIONS:
Device: Duodena-jejunal liner
  Other Names: Endobarrier
  Arms: Duodeno - jejunal liner

SUMMARY:
Obesity and its complications have a significant effect on morbidity and mortality in these subjects. Especially at risk are subjects with extremely increased BMI (above 99th percentile for age and gender in adolescents). In these subjects classical treatment with diet and cognitive therapy has a limited effect. Bariatric procedures, at the moment, are the only feasible therapeutic possibility.

Bariatric procedures are based on several principles; restrictive, malabsorptive and combined. They can be surgical or endoscopic. The later are used in subjects that do not qualify for surgical procedures that decline them or are used before a planed definite bariatric procedure.

Duodena-jejunal liner (DJL) is an endoscopic tool, that is efficiently and safely used to decrease body weight and ameliorated obesity complications, especially those associated with diabetic state.

Aims of the study are:

* To determine (short and long-term) efficacy of DJL in decreasing body weight in adolescents.
* To determine (short and long-term) efficacy of DJL in ameliorating complications of morbid obesity - abnormal glucose metabolism, dislipidemia, altered adipokine secretion pattern, altered secretion pattern of gastrointestinal hormones in adolescents.
* To visualize functional alternations in the selected central nervous system regions associated with appetite regulation upon insertion of DJL.
* To evaluate psychological outcomes; change in emotional and behaviour problems, in body image, in eating disorder symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Subjects estimated to fully comply with study protocol and have signed an informed consent form.
* Age > 15 years.
* BMI ≥ 99. percentile for age and gender.
* Inefficient conservative measures (of at least 6 months duration) to decrease body weight (characterized as a decrease in BMI > 10 %).
* Documented negative pregnancy test in women of childbearing potential.
* Women of childbearing potential agree to remain on contraceptives for the duration of their trial participation.

Exclusion Criteria:

* Previous GI surgery that could potentially affect the ability to place sleeve or affect the function of the implant.
* Subjects with congenital or acquired anomalies of the GI tract which in the opinion of the investigator, may impair implantation of the EndoBarrier device.
* Subjects who had gastrooesophageal reflucs disease..
* Known abnormal pathologies or conditions of the gastrointestinal tract, including ulcers or Crohn's disease, upper gastro-intestinal bleeding conditions.
* Coagulopathy defined as Hgb <10g/dl and platelet < 100,000/ml or diagnosis of other severe coagulopathy like hemophilia.
* Any documented history of acute or chronic pancreatitis.
* Subjects requiring regular antithrombotic therapy (i.e. anticoagulant or antiplatelet agent).
* Known diagnosis of systemic lupus erythematosus, scleroderma or other autoimmune connective tissue disorder.
* Subject is or has been enrolled in another investigational study within 6 months of participation into the EndoBarrier study.
* Subjects who are mentally retarded or emotionally unstable.
* Subjects who are pregnant or were breastfeeding.
* Subjects with an abnormal laboratory or ECG abnormality which the investigators deems clinically significant and makes the patient a poor candidate for the study.

Ages: 16 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 22 (Actual)
Dates: Start 2014-07; Primary Completion 2018-12-10 (Actual); Study Completion 2018-12-20 (Actual)

PRIMARY OUTCOMES:
Change in BMI (BMI SDS) | 12 and 24 months

SECONDARY OUTCOMES:
Change in basal and stimulated glucose and insulin levels | 12 and 24 months
Change in cholesterol levels | 12 and 24 months
Change in selected gut hormones | 12 and 24 months
Change in selected adipokine and inflammatory cytokines levels | 12 and 24 months
Change in activity of selected appetite-associated central nervous system regions. | 12 and 24 months
Change in emotional and behaviour problems, body image and eating disorder symptoms | 12 and 24 months

OTHER OUTCOMES:
Safety profile of DJL in adolescents. | 12 months
  Number of participants with adverse events (pain, nausea, vomiting, bleeding, gastrointestinal obstruction) and number of adverse events will be used to measure safety and tolerability of the investigated device in adolescents.

CONTACTS AND LOCATIONS:
Overall Officials: Tadej Battelino, MD, PhD, Principal Investigator — UMC Ljubljana
Locations (1):
- UMC Ljubljana, Ljubljana, Slovenia

REFERENCES:
- [Background] Escalona A, Pimentel F, Sharp A, Becerra P, Slako M, Turiel D, Munoz R, Bambs C, Guzman S, Ibanez L, Gersin K. Weight loss and metabolic improvement in morbidly obese subjects implanted for 1 year with an endoscopic duodenal-jejunal bypass liner. Ann Surg. 2012 Jun;255(6):1080-5. doi: 10.1097/SLA.0b013e31825498c4. PMID 22534421
- [Background] de Moura EG, Martins BC, Lopes GS, Orso IR, de Oliveira SL, Galvao Neto MP, Santo MA, Sakai P, Ramos AC, Garrido Junior AB, Mancini MC, Halpern A, Cecconello I. Metabolic improvements in obese type 2 diabetes subjects implanted for 1 year with an endoscopically deployed duodenal-jejunal bypass liner. Diabetes Technol Ther. 2012 Feb;14(2):183-9. doi: 10.1089/dia.2011.0152. Epub 2011 Sep 20. PMID 21932999
- [Background] de Moura EG, Orso IR, Martins BC, Lopes GS, de Oliveira SL, Galvao-Neto Mdos P, Mancini MC, Santo MA, Sakai P, Ramos AC, Garrido-Junior AB, Halpern A, Cecconello I. Improvement of insulin resistance and reduction of cardiovascular risk among obese patients with type 2 diabetes with the duodenojejunal bypass liner. Obes Surg. 2011 Jul;21(7):941-7. doi: 10.1007/s11695-011-0387-0. PMID 21442376